CLINICAL TRIAL: NCT04627233
Title: The Clinical Trial of Application of Ezrin Peptide (HEP-1) for Treatment of Coronavirus Disease (COVID-19) Infection
Brief Title: Ezrin Peptide (HEP-1) for Treatment of Coronavirus Disease (COVID-19) Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: praxisgemeinschaft für zelltherapie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SBMU.REC.1399.023
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Treatment; Corona Virus Infection
Keywords: COVID19; Treatment; Ezrin peptide; HEP-1
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention:control group (Placebo Comparator)
  Interventions: Drug: Placebo
- Experimental:Intervention group (Experimental)
  Interventions: Drug: Human Ezrin Peptide 1 (HEP1)

INTERVENTIONS:
Drug: Human Ezrin Peptide 1 (HEP1) — HEP-1 will be administrated s.c. into the lower abdominal wall
  1. induction dosage: 2 mg Ezrin in 2 ml physiological saline applied s.c.,one injection every 12 hours until symptoms disappear followed by
  2. maintenance dosage: 0.2 mg Ezrin in 1 ml physiological saline solution s.c 1/day for 10 days
  Arms: Experimental:Intervention group
Drug: Placebo — placebo group received normal saline in a same volume to match corresponding HEP-1 doses. Study drug was administered by qualified staff in research clinic settings; injections were given to abdominal sites on rotating basis, by anatomic quadrant.
  Arms: No intervention:control group

SUMMARY:
Currently, SARS-CoV-2 the novel member of the corona virus family, affecting the world leading to COVID-19 disease. It can result life-threatening condition by developing severe acute respiratory distress syndrome (ARDS). Based on previous evidence a group of patients with severe COVID-19 develop a cytokine storm syndrome which leads to hyper-inflammation lung tissue damage. Supportive care is the current management of COVID-19 is and management of ARDS as a main cause of mortality has been remained challenging. Therefore, an urgent effective treatment of COVID-19 regarding hyper-inflammation mechanism is required. Currently, development of novel anti-viral agents and vaccines are the main issues. However, it needs long time, from months to years, until suitable new medications and vaccines have been developed. An immune-modulatory tetra deca peptide (14-mer peptide) named Human Ezrin Peptide 1 (HEP-1) (trade name Gepon) was introduced by the group of Ataullakhanov in Russia. Regarding its proved anti-viral and anti-inflammatory effect, Russian authorities approved Gepon for treatment of ulcerative colitis treatment and Hepatitis -C.

In this regard, it seems that Hep-1 is a very safe immune-modulatory agent which can be effective in the management of COVID-19 infection without any adverse effect for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with a positive SARS-CoV-2 PCR test and presenting with one or more clear clinical symptoms of COVID-19 disease
* No contraindication to HEP-1
* Obtained informed consent

Exclusion Criteria:

* Patients who had received any immuno-modulator therapy
* Active or chronic kidney/ liver diseases,
* Oncological diseases
* Other viral infection including HIV and hepatitis.
* Any allergic reaction or sensitivity to HEP-1
* Breast feeding or pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-12-20 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to clinical improvement of disease symptoms | 7 days
Duration of Hospitalization | 28 days
Duration of artificial ventilation | 28 days

SECONDARY OUTCOMES:
CT Severity score | 28 days
  Range 0-40
CBC | 28 days
IL-1 | 28 days
IL-6 | 28 days
TNF | 28 days
CRP | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shahid Beheshti University of Medical Sciences, Tehran, Iran

REFERENCES:
- [Background] Bretscher A, Reczek D, Berryman M. Ezrin: a protein requiring conformational activation to link microfilaments to the plasma membrane in the assembly of cell surface structures. J Cell Sci. 1997 Dec;110 ( Pt 24):3011-8. doi: 10.1242/jcs.110.24.3011. PMID 9365271
- [Background] Pore D, Gupta N. The ezrin-radixin-moesin family of proteins in the regulation of B-cell immune response. Crit Rev Immunol. 2015;35(1):15-31. doi: 10.1615/critrevimmunol.2015012327. PMID 25746045
- [Background] Pore D, Parameswaran N, Matsui K, Stone MB, Saotome I, McClatchey AI, Veatch SL, Gupta N. Ezrin tunes the magnitude of humoral immunity. J Immunol. 2013 Oct 15;191(8):4048-58. doi: 10.4049/jimmunol.1301315. Epub 2013 Sep 16. PMID 24043890
- [Background] Millet JK, Kien F, Cheung CY, Siu YL, Chan WL, Li H, Leung HL, Jaume M, Bruzzone R, Peiris JS, Altmeyer RM, Nal B. Ezrin interacts with the SARS coronavirus Spike protein and restrains infection at the entry stage. PLoS One. 2012;7(11):e49566. doi: 10.1371/journal.pone.0049566. Epub 2012 Nov 21. PMID 23185364